CLINICAL TRIAL: NCT00953953
Title: Study of the Phenomenon of Dynamic Left Ventricular Dyssynchrony in Heart Failure Patients and Its Clinical Significance.
Brief Title: Study of Left Ventricular Dyssynchrony in Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Darshak Karia, MD, Director, Heart Failure Services, Albert Einstein Healthcare Network
Other Study IDs: HN 3052
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Acutely Decompensated Systolic HF: Patients with moderate or severe Heart Failure (defined ast NYHA class III or IV).
  Interventions: Device: Phillips ultrasound system
- Chronic HF Patients on Dialysis: Patients who have heart failure (defined as NYHA class II, III, or IV) and are on dialysis.
  Interventions: Device: Phillips ultrasound system
- Ambulary Chronic HF: Patients with diagnosis of chronic heart failure (NYHA class II and III) who are on optimal medical therapy.
  Interventions: Device: Phillips ultrasound system
- Acutely Decompensated Diastolic HF: Patients with moderate or severe Heart Failure (defined ast NYHA class III or IV).
  Interventions: Device: Phillips ultrasound system

INTERVENTIONS:
Device: Phillips ultrasound system — The tissue doppler imaging color images will be acquired from two, three, and four-chamber apical views to assess the longitudinal contraction of the left ventricle.

SUMMARY:
Heart failure has become one of the major epidemics of the modern era. Despite optimal standard drug therapy, the prognosis of patients with heart failure remains poor. Patient with Heart Failure are prone to have "dyssynchrony" which means that there are electrical disturbances that cause the heart to pump blood in an inefficient way. Ventricular dyssynchrony has been associated with increased mortality in patients with heart failure. Based on these observations, techniques have been developed to correct dyssynchrony. The investigators propose to investigate the change of dyssynchrony in relation to intravascular volume status and exercise in heart failure patients. The investigators also propose to examine dyssynchrony in the setting of acutely decompensated heart failure. The change in dyssynchrony will be followed to examine if it translates into clinical significance.

DETAILED DESCRIPTION:
Heart failure has become one of the major epidemics of the modern era. Despite optimal standard drug therapy, the prognosis of patients with heart failure remains poor. It has been noted that 15% of all HF patients and 30% of those with NYHA class III and IV HF have intraventricular conduction delay, with a QRS duration >120 ms, most commonly manifested as LBBB. These electrical disturbances result in LV dyssynchrony, seen as a paradoxical septal wall motion activity, suboptimal ventricular filling and mitral regurgitation; thus further compromising an already dysfunctioning left ventricle. Ventricular dyssynchrony has been associated with increased mortality in patients with heart failure.

Based on these observations, techniques have been developed to correct dyssynchrony. Cardiac resynchronization therapy (CRT) has been shown to improve subjective and objective parameters in heart failure patients with QRS duration > 120msec. However, there is a group of heart failure patients who did not respond to CRT. Also it has been noted that approximately 30% of heart failure patients with QRS duration > 120 msec do not have actual mechanical dyssynchrony by tissue doppler imaging. The electromechanical discrepancy of ventricular dyssynchrony has been suggested as the possible explanation for the lack of response. Also, there are heart failure patients with normal QRS duration who do have mechanical dyssynchrony. These findings bring more emphasis to the importance of mechanical dyssynchrony than electrical dyssynchrony, which is measured by QRS duration on surface EKG.

There are many different modalities to quantify mechanical dyssynchrony. The most commonly used method is tissue doppler imaging (TDI). TDI measures the velocities of myocardial tissue and time to maximal velocities. Then, these are used to describe contractions of different wall segments. Strain and strain rates are more sophisticated ways to measure active segment contraction rather than passive movements.

We propose to investigate the change of dyssynchrony in relation to intravascular volume status and exercise in heart failure patients. We also propose to examine dyssynchrony in the setting of acutely decompensated heart failure. The change in dyssynchrony will be followed to examine if it translates into clinical significance.

ELIGIBILITY:
ACUTELY DECOMPENSATED SYSTOLIC HEART FAILURE

Inclusion Criteria:

* Patients over the age of 18 and able to consent
* NYHA Class III or IV
* EF≤ 35%
* Diagnosis of acute congestive heart failure exacerbation by history or physical examination
* Ability to understand and willing to sign informed consent
* Willingness to follow-up for clinic visits at 30 days and 6 months

Exclusion Criteria:

* Pacemaker
* Patients requiring and willing to sign informed consent
* Unwillingness to provide consent

CHRONIC HEART FAILURE on DIALYSIS GROUP

Inclusion Criteria:

* Patients over the age of 18 and able to consent
* NYHA Class II, III, or IV
* EF ≤ 35% with a screening echocardiogram
* Ability to understand and willing to sign informed consent
* Willingness to follow up at 30 days and 6 months via phone contact

Exclusion Criteria:

* Unwillingness to provide consent
* Pacemaker

AMBULATORY CHRONIC HEART FAILURE GROUP

Inclusion Criteria:

* Patients over the age of 18 and able to consent
* NYHA Class II and III with an EF ≤ 35%
* Diagnosis of chronic heart failure and currently on optimal medical therapy, including ACE, or ARB, beta-blockers and diuretics including spironolactone
* Ability to understand and willing to sign informed consent
* Willingness to follow up as an outpatient at 30 days and 6 months

Exclusion Criteria:

* Incapable of taking the 6-minute walk test due to any condition unrelated to heart failure
* Patients requiring chronic inotrope therapy
* Pacemaker
* Symptoms of angina limiting exercise ability
* Unwillingness to provide consent

ACUTELY DECOMPENSATED DIASTOLIC HEART FAILURE GROUP

Inclusion Criteria:

* Patients over the age of 18 and able to consent
* NYHA Class III or IV
* EF ≥ 45%
* Diagnosis of acute congestive heart failure exacerbation by history or physical examination
* Ability to understand and willing to sign informed consent
* Willingness to follow-up for clinic visits at 30 days and 6 months

Exclusion Criteria:

* Pacemaker
* Patients requiring inotrope support on admission
* Unwillingness to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely Decompensated Systolic HF group: patients who are admitted to Albert Einstein Medical Center on the HF service.
  Chronic HF on Dialysis group: patients at the dialysis center at Albert Einstein Medical Center.
  Ambulatory Chronic HF group: patients who present to the Albert Einstein Medical Center HF clinic.
  Acutely Decompensated Diastolic HF group: patients who are admitted to Albert Einstein Medical Center on the HF service.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Acutely Decompensated Systolic HF Group:Assess the incidence of change in dyssynchrony at admission and prior to discharge during acute decompensated heart failure exacerbation hospitalization | 6 months
Chronic Heart Failure on Dialysis Group: Assess the incidence of change in dyssynchrony before, during, and after dialysis | 6 months
Ambulatory Chronic Heart Failure Patients Group: Assess the incidence of change in dyssynchrony at rest and during peak exercise in Chronic Heart failure patients. | 6 months
Acutely Decompensated Diastolic Heart Failure Group: Assess the incidence of change in dyssynchrony at admission and prior to discharge during acutely decompensated diastolic heart failure exacerbation hospitalization | 6 months

SECONDARY OUTCOMES:
All four arms: Determine the change of dyssynchrony | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Darshak Karia, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States